CLINICAL TRIAL: NCT01925703
Title: Short-Term Effects & Safety of an Accelerated Intravenous Iron Regimen in Patients With Heart Failure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-0551
Record Dates: First submitted 2013-05-30; First posted 2013-08-20 (Estimated); Results first posted 2015-08-10 (Estimated); Last update posted 2015-08-25 (Estimated); Status verified 2014-05

CONDITIONS: Heart Failure; Iron Deficiency Anemia
MeSH Terms: conditions — Heart Failure; Anemia, Iron-Deficiency | interventions — ferric gluconate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sodium ferric gluconate (Experimental): Sodium ferric gluconate 250 mg administered intravenously every 12 hours until iron repletion completed (as determined by Ganzoni equation) or patient discharge, whichever comes first.
  Interventions: Drug: Sodium ferric gluconate

INTERVENTIONS:
Drug: Sodium ferric gluconate — Sodium ferric gluconate 250 mg administered intravenously every 12 hours until iron repletion completed (as determined by Ganzoni equation) or patient discharge, whichever comes first.
  Other Names: Ferrlecit

SUMMARY:
Intravenous iron replacement has been shown to benefit patients with heart failure and iron deficiency, but the weekly outpatient regimens studied to date are impractical for many patients. Our purpose is to evaluate the short-term effects and safety of an accelerated intravenous iron regimen in hospitalized patients with these two conditions.

DETAILED DESCRIPTION:
The purpose of this pilot investigation is to evaluate the short-term hematologic effects and safety of an accelerated intravenous iron regimen in patients with heart failure and iron deficiency. Recent investigations have demonstrated improved clinical outcomes with the use of intravenous iron therapy in this patient population, but a weekly regimen administered to ambulatory patients may be inconvenient, impractical, and associated with less than optimal adherence rates for many patients, especially those with reduced functional capacity. The heart failure population is characterized by frequent hospitalizations, which would make an accelerated inpatient regimen a convenient and attractive option for improving heart failure symptoms, exercise tolerance, and quality of life. Accelerated regimens have been demonstrated as being both safe and effective in other patient populations, but no studies to date have evaluated this strategy in hospitalized patients with heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Admission to the general cardiology or heart failure services and under the care of a cardiologist at the study institution
* New York Heart Association Class II-IV heart failure
* Ejection fraction < 40%
* Serum hemoglobin < 12.0 g/dL
* Ferritin < 100 ng/mL or 100-300 ng/mL with transferrin saturation (TSAT) < 20%
* Patients deemed by an attending physician to require intravenous iron therapy based on previous attempts to correct iron deficiency or other patient-specific circumstances

Exclusion Criteria:

* Anemia of other known etiology (e.g., malignancy, malabsorption syndromes)
* Use of iron or erythropoietin-stimulating agents within previous 12 weeks
* Blood transfusion within previous 12 weeks; additionally, if patients receive blood transfusions during the study period, they will remain in the safety analysis but will be excluded from efficacy analysis
* Active bleeding
* Known infection at admission
* Immunosuppressant therapy
* Renal replacement therapy
* Known pregnancy
* Any other criteria deemed by the attending physician to warrant exclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2011-04; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jo Ellen Rodgers, PharmD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina Hospitals & Clinics, Chapel Hill, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sodium Ferric Gluconate
Started | 13
Dosing Regimen Completed | 12
Full Iron Repletion Achieved | 11
Follow-up Completed | 9
Completed | 9
Not Completed | 4
Not completed — Physician Decision | 1
Not completed — Lost to Follow-up | 2
Not completed — Discharge prior to full iron repletion | 1

BASELINE CHARACTERISTICS:
Arm/Group | Sodium Ferric Gluconate
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.9 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 13
Weight [Mean (Standard Deviation); unit: kilograms] | 94.9 (25)
Body Mass Index [Mean (Standard Deviation); unit: kilograms per meter squared] | 33.9 (9.5)
NYHA Heart Failure Class [Number; unit: participants]
  Class I | 0
  Class II | 0
  Class III | 7
  Class IV | 6
Ejection Fraction [Mean (Standard Deviation); unit: percent] | 20.2 (8.4)
Hemoglobin Concentration [Mean (Standard Deviation); unit: grams per deciliter] | 10.6 (1.4)
Ferritin Concentration [Mean (Standard Deviation); unit: nanograms per milliliter] | 86.4 (61.4)
Transferrin Saturation [Mean (Standard Deviation); unit: percentage of transferrin saturation] | 11.7 (4.6)
Serum Creatinine Concentration [Mean (Standard Deviation); unit: milligrams per deciliter] | 1.2 (0.4)

OUTCOME MEASURES:

1. Primary Outcome: Serum Hemoglobin Concentration
Description: Change in serum hemoglobin concentration compared to baseline and at follow-up within 1-4 weeks after last intravenous iron infusion
Time Frame: Baseline and at follow-up within 1-4 weeks
Population: All patients who achieved complete iron repletion for whom follow up data were available.
Measure: Mean (95% Confidence Interval); unit: grams per deciliter
Arm/Group | Sodium Ferric Gluconate
Number analyzed (Participants) | 9
grams per deciliter | 1.2 [0.45 to 1.9]

2. Secondary Outcome: Transferrin Saturation
Description: Change in transferrin saturation compared to baseline and at follow-up within 1-4 weeks after last intravenous iron infusion
Time Frame: Baseline and at follow-up within 1-4 weeks
Population: All patients who achieved complete iron repletion for whom follow-up data were available.
Measure: Mean (95% Confidence Interval); unit: Percentage of transferrin saturation
Arm/Group | Sodium Ferric Gluconate
Number analyzed (Participants) | 9
Percentage of transferrin saturation | 10.5 [6.5 to 14.6]

3. Secondary Outcome: Serum Ferritin Level
Description: Change in serum ferritin level compared to baseline and at follow-up within 1-4 weeks after last intravenous iron infusion
Time Frame: Baseline and at follow-up within 1-4 weeks
Population: All participants who achieved complete iron repletion for whom follow up data were available.
Measure: Mean (95% Confidence Interval); unit: nanograms per milliliter
Arm/Group | Sodium Ferric Gluconate
Number analyzed (Participants) | 9
nanograms per milliliter | 364.2 [129.7 to 598.7]

ADVERSE EVENTS:
Arm/Group | Sodium Ferric Gluconate
Serious Adverse Events (participants affected / at risk) | 1/13
Other Adverse Events (participants affected / at risk) | 11/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sodium Ferric Gluconate (N=13)
Clinical Deterioration (General disorders) | 1 (1) — Patient was withdrawn from study after two of the four study drug doses were administered at the discretion of the treating physician. Reason for withdrawal was clinical deterioration secondary to hypovolemia and aggressive vasodilator titration.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sodium Ferric Gluconate (N=13)
nausea (Gastrointestinal disorders) | 3 (6)
constipation (Gastrointestinal disorders) | 1 (1)
abdominal discomfort (Gastrointestinal disorders) | 3 (5)
diarrhea (Gastrointestinal disorders) | 3 (4)
injection site itching (Skin and subcutaneous tissue disorders) | 3 (3)
injection site discomfort (Skin and subcutaneous tissue disorders) | 3 (4)
thrombophlebitis (Vascular disorders) | 1 (1)
cellulitis (Skin and subcutaneous tissue disorders) | 1 (1)
headache (Nervous system disorders) | 2 (2)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
leg cramps (Musculoskeletal and connective tissue disorders) | 1 (1)
bladder discomfort (Renal and urinary disorders) | 1 (1)
fatigue (General disorders) | 1 (1)
chills (General disorders) | 1 (1)
melena (Gastrointestinal disorders) | 1 (1)
hematuria (Renal and urinary disorders) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No